CLINICAL TRIAL: NCT02524496
Title: Limited Access, Open-label, Compassionate Use of Cisapride in the Treatment of Gastroparesis
Brief Title: Limited Access Protocol for the Use of Oral Cisapride
Status: Completed | Type: Observational
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Other Study IDs: 0009012025
Record Dates: First submitted 2007-12-25; First posted 2015-08-14 (Estimated); Last update posted 2015-08-14 (Estimated); Status verified 2015-08

CONDITIONS: Gastroparesis
MeSH Terms: conditions — Gastroparesis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Due to the lack of other drugs to treat gastroparesis Janssen and FDA approved the compassionate use of cisapride to treat patients who had no other effective therapy. For this observational study, 3 patients who had already been prescribed cisapride by outside physicians, were followed to determine the effectiveness of cisapride on their gastric emtpying.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of gastroparesis.

Exclusion Criteria:

* No diagnosis of gastroparesis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The subjects of the study were diagonosed with gastroparesis that was not being adequately treated.
Sampling Method: Non-Probability Sample
Enrollment: 3 (Actual)
Dates: Start 2001-03; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Improvement in gastric emptying via self-report | ten years
  Patients were asked at clinical appointments about problems and improvement with gastric emptying.